CLINICAL TRIAL: NCT03113799
Title: A Study to Evaluate the Performance and Safety of Aqueduct's Smart External Device (SED) Compared to Standard EVD Drains
Brief Title: A Study Evaluate Aqueduct's Smart External Drain
Acronym: SED
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aqueduct Critical Care (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ASSESSED SED1
Record Dates: First submitted 2017-03-20; First posted 2017-04-14 (Actual); Last update posted 2019-01-31 (Actual); Status verified 2019-01

CONDITIONS: Hydrocephalus; Hydrocephalus in Children; Tumor, Brain
MeSH Terms: conditions — Hydrocephalus; Brain Neoplasms

STUDY DESIGN:
Intervention Model Description: In this study the subject will act as their own control and will be treated on day one with the standard of care EVD and then on Day 2 treated with the SED.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Single Arm study (Other): Single Arm study In this study, the subject will act as their own control. On Day 1 of the two day study, the subject will be observed while treated on their standard EVD. On Day 2, the subject will be treated with the Smart External Drain (SED).
  Interventions: Device: Smart External Drain - SED

INTERVENTIONS:
Device: Smart External Drain - SED — Subject will be treated on Day 2 with the SED. ICP and CSF volumes will be recorded at prespecified intervals while subject is stationary and while subject is engaged in protocol-driven directed movements.

SUMMARY:
To evaluate the performance characteristics of the Smart External Drain (SED) compared with standard EVD drains in the hospital setting, specifically:

* Number, type and duration of staff interactions.
* Regulating and controlling ICP and CSF drainage.
* Maintaining system control with patient movement.

DETAILED DESCRIPTION:
In this two day clinical trial, subjects will be observed on Day 1 of study during their routine treatment and using their already existing EVD. On Day 2 of study; subjects will be switched to the Smart External Drain for monitoring and management of ICP and CSF

ELIGIBILITY:
Inclusion Criteria:

1. Stable Neuro - examination on standard EVD assessed as Not Clinically Significant (NCS) by PI or delegated Sub-I prior to study treatment.
2. GCS > 13 (minimum of E3V5M5) prior to study treatment.
3. Subject must be scheduled to have an EVD placed as part of routine management and for a length of at least 48 hours. (e.g. in the setting of a tumor removal or treatment of hydrocephalus)
4. Age 5-80.
5. Stable Vital Signs - Blood pressure (Systolic and Diastolic), Heart Rate, Respiratory Rate and weight assessed as not clinically significant (NCS) and afebrile as per PI/Sub-assessment. (Stable Vital signs will be re-assessed again prior to treatment with the SED on Day 2)
6. Able to perform and follow simple commands (ex: sit up in bed, lay down in bed)
7. Pre-Study CT/MRI Imaging stable per PI Sub-I Assessment post ventriculostomy.
8. Able to stand
9. Able to obtain consent

Exclusion Criteria:

1. Refractory ICP or needing active ICP management
2. Unable to tolerate brief clamping of EVD (<5min)
3. Unable to follow simple commands
4. Unconscious
5. Anticoagulant Therapy
6. Known bleeding diathesis
7. Scalp Infection
8. In the opinion of the Investigator the subject is not a good study candidate

Ages: 5 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2017-04-12 (Actual); Primary Completion 2018-08-15 (Actual); Study Completion 2019-01-29 (Actual)

PRIMARY OUTCOMES:
Staff interactions | Two Days
  Average number of staff interactions per patient with standard EVD compared to intervention, the Smart External Drain (SED)

SECONDARY OUTCOMES:
Staff Time | Two Days
  Total minutes spent by staff interacting with standard EVD compared to SED
Safety | Two Days
  Number of Participants with Adverse Events That Are Related to Treatment

CONTACTS AND LOCATIONS:
Overall Officials: Sam Browd, MD, PhD, Study Director — Aqueduct Critical Care, Inc
Locations (2):
- United States (2):
  - Seattle Children's Hospital, Seattle, Washington
  - University of Washington School of Medicine / Harborview Medical Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Undecided